CLINICAL TRIAL: NCT02677402
Title: Effects of Thermo Neutral Water Immersion, Cold-water Immersion and Contrast Water Therapy on Lower Limb Veins Calibres
Brief Title: Effects of Various Modalities Water Immersion on Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Franche-Comté (Other)
Responsible Party: Principal Investigator, Laurent Mourot, PhD, University of Franche-Comté
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H2O
Record Dates: First submitted 2016-01-10; First posted 2016-02-09 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hydrotherapy
Keywords: femoral vein; saphenous vein; hydrostatic pressure; temperature; recovery
MeSH Terms: interventions — Immersion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cold water immersion (Experimental): Participants immersed their lower limbs in water of ~12°C
  Interventions: Other: immersion
- contrast water therapy (Experimental): Participants immersed their lower limbs in water : alternated every 2 min between ~12°C and ~35°C for CWT
  Interventions: Other: immersion
- thermo neutral immersion (Experimental): Participants immersed their lower limbs in water of ~35°C
  Interventions: Other: immersion

INTERVENTIONS:
Other: immersion

SUMMARY:
Objectives In this study the investigators examined the changes in common femoral vein (CFV) and great saphenous vein (GSV) calibre during thermo neutral water immersion (TNI), cold water immersion (CWI) and contrast water therapy (CWT).

Design Ten professional handball players visited the laboratory on three occasions. At each visit, participants completed a 20-minutes procedure in an upright position: 4-minutes in air (baseline) and then 16-minutes lower limbs TNI (~35°C), CWI (~12°C) or CWT (2:2minutes (~12°C to ~35°C) ratio), selected randomly.

Methods CFV and GVS calibres were evaluated by echo Doppler measures at baseline and at the end of 16 min immersion.

ELIGIBILITY:
Inclusion Criteria:

* Free healthy voluntary

Exclusion Criteria:

* hypersensitivity to cold

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
change in common femoral vein cross-section (mm2) during three immersion modalities immersion | Change from Baseline at 16 min of immersion in 3 modalities, doppler ultrasound measurements
  thermo neutral water immersion (TNI), cold water immersion (CWI) and contrast water therapy (CWT)
change in great saphenous vein antero posterior diameter (mm) during three immersion modalities immersion | Baseline at 16 min of immersion in 3 modalities, doppler ultrasound measurements
  thermo neutral water immersion (TNI), cold water immersion (CWI) and contrast water therapy (CWT)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Beliard, MD, Principal Investigator — University of Franche-Comte
Locations (1):
- Beliard, Besançon, France

IPD SHARING:
Plan to Share IPD: No